CLINICAL TRIAL: NCT02794116
Title: Survival of Sealants in Molars Affected by Molar-Incisor Hypomineralization
Brief Title: Sealants in Molars Affected by Molar-Incisor Hypomineralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Juliana Feltrin de Souza Caparroz, Professor, Universidade Federal do Paraná
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFParana_1
Record Dates: First submitted 2016-05-02; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group: Sound teeth (Active Comparator): 20 first permanent molars sound, that not affected by MIH will be included.
  The teeth were treated with conventional sealants to prevent caries lesion
  Interventions: Procedure: Conventional Sealants
- Test: Hypomineralized teeth (Experimental): 20 first permanent molars affected by MIH will be included.
  The MIH teeth were treated with a resin sealants.
  Interventions: Procedure: Resin Sealants

INTERVENTIONS:
Procedure: Conventional Sealants — It is a preventive treatment for caries lesions. The procedure following operative sequence: prophylaxis; absolute isolation; application of 37.5% phosphoric acid for 30 s in enamel; extensive washing; drying with cotton and air jet for 5 s; sealing with resin sealant application (Fluroshield, NY, USA), according to manufacturer guidelines; removal absolute isolation; examination of occlusal contact and final polishing.
  Other Names: Control group
  Arms: Control group: Sound teeth
Procedure: Resin Sealants — It is a resin sealants to preventive treatment for caries lesions. The procedure following operative sequence: prophylaxis; absolute isolation; application of 37.5% phosphoric acid for 30 s in enamel; extensive washing; drying with cotton and air jet for 5 s; sealing with resin sealant application (Fluroshield, NY, USA), according to manufacturer guidelines; removal absolute isolation; examination of occlusal contact and final polishing.
  Other Names: Test group
  Arms: Test: Hypomineralized teeth

SUMMARY:
Aim: To evaluate the clinical survival of fluoride sealants applied in first permanent molars affected by Molar-Incisor Hypomineralization (MIH).

Material and Methods: For this case control study, it was selected 41 first permanent molars of the 21 children aged 6-8 years. MIH was classified by one calibrated examiner (kappa 0.80) according severity of the MIH lesion (EAPD, 2003). Inclusion criteria were FPM with MIH or sound (without MIH), fully erupted, and with sealant treatment indication.

The FPMs were assigned into two groups: G1 - Control group and G2 - MIH group. Both group teeth were treated with sealant application (Fluroshield, NY, USA). Clinical follow-up was performed at baseline, 1, 6, 12 and 18 months for anatomic form, marginal adaptation, retention and presence of caries, according to the United States Public Health Service USPHS-Modified by a blinded examiner (kappa 0.80). The Acturial Method was used to evaluate the survival of sealants. Statistical analysis compared the ratings of each criterion between materials using the Fisher's exact test at a level of significance of 5% (p<0.05).

DETAILED DESCRIPTION:
This study was conducted according to the Helsink Declaration. The approval was obtained from the Ethics and Research Committee at Araraquara Dental School, São Paulo, Brazil (protocol #11/09). All parents/guardians of the children signed the informed consent.

Study design:

This case control study included four clinical exams performed in 6 to 8 years-old children that received preventive treated with sealants, divided into 2 groups: G1 - teeth not affect by MIH and G2 - teeth affect by MIH.

Subjects:

The 21 children included in the study had been previously diagnosed with MIH, according to the EAPD criteria. A total of 41 first permanent molars teeth (FPM) were included, being 16 without MIH and 25 with MIH.

Calibration of the examiner for the evaluations:

The examiner was calibrated according to MIH based on criteria proposed by the European Academy of Pediatric Dentistry and for USPHS-Modified. The examiner assessed 32 clinical photographs of patients from the Clinic of Pediatric Dentistry of the Araraquara Dental School in São Paulo, Brazil, followed by a discussion with the MIH research team of all the indices and codes. After an agreement, 30 patients with enamel alterations (17 of them with MIH) were evaluated. After 2 weeks, the patients were reevaluated and the Kappa coefficient was used to verify the agreement between the evaluations. The intra-examiner values for MIH and USPHS-modified were 0.80.

Treatment:

The 41 FMP were clinically examined and classified according the presence of MIH according the European Association of Paediatric Dentistry and were distributed into groups. The preventive procedures were performed at the Pedodontics Clinics of São Paulo State University, for another operator. All teeth receive pre-treat with care 4 weekly applications of fluoride varnish (Duraphat, NY, USA).

Both group teeth were treated with sealants.

Evaluation:

The four clinical exams (1, 6, 12 and 18 months) were performed in a clinical environment according exams preconized by the World Health Organization under artificial lights and after prophylaxis.

The sealants were clinically evaluated by a calibrated examiner (Kappa 0.80). The groups were evaluated according to the criteria for quality of the restoration proposed by the United States Public Health Service USPHS-Modified and classified as satisfactory or unsatisfactory. When the tooth was considered unsatisfactory, it was considered failure and the treatment was replaced but it had not considered for the research evaluations.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were children born and living in Araraquara/SP (Brazil), 6 to 8-year-aged, presenting FPM with MIH or sound, fully erupted, with sealant treatment indication.

Exclusion Criteria:

* It was excluded teeth with enamel breakdown, enamel tooth malformation linked to syndromes, dental fluorosis, amelogenesis imperfect, fixed orthodontic appliances and patients with bruxism.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
clinical Survival of the sealants | 6 months
  The sealants were assessed using the according to the United States Public Health Service-Modified criteria, which the data were analyzed in scores
clinical survival of the sealants | 18 months
  The sealants were assessed using the according to the United States Public Health Service-Modified criteria, which the data were analyzed in scores

IPD SHARING:
Plan to Share IPD: Yes